CLINICAL TRIAL: NCT03801447
Title: Ratio of Angiogenesis-related Biomarkers (sFlt-1/PlGF) in the Prediction Of mateRnal & feTal outcomeS
Brief Title: Biomarkers and Preeclampsia Outcomes
Acronym: REPORTS
Status: Completed | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Maternity Center of Tunis (Unknown)
Responsible Party: Sponsor
Other Study IDs: DAC-003-REPORTS
Record Dates: First submitted 2018-05-27; First posted 2019-01-11 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, observational, monocentric, non-interventional study.

DETAILED DESCRIPTION:
In practice, patients with preeclampsia are referred to the hospital for medical management only clinical signs & symptoms and standard biological tests are available for patient individualized care. Hence, a new diagnostic tool to distinguish and stratify the different patients referred is in need of proper triage.

REPORTS study aims to determine the diagnostic utility of 2 preeclampsia biomarkers (sFlt-1/PlGF ratio) in clinical decision making in preeclamptic women.

Data are collected by DACIMA Clinical Suite, according to FDA 21 CFR part 11 requirements (Food and Drug Administration 21 Code of Federal Regulations part 11), the HIPAA specifications (Health Insurance Portability and Accountability Act), and the ICH standards (International Conference on Harmonisation)

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed preeclampsia
* Singleton pregnancy
* Between 26 weeks of gestation and 37 weeks of gestation & 6 days

Exclusion Criteria:

* Multiple pregnancies

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Preeclampsia was defined according to the ACOG (The American College of Obstetricians and Gynecologists). The diagnosis of Preeclampsia was based on clinical judgment and routine laboratory findings at inclusion.
  Patients were suspected of Preeclampsia if they:
  * presented with new onset hypertension and or proteinuria at or after 20 weeks of gestation
  * developed an aggravation of their preexisting hypertension and or preexisting proteinuria
  * or if they presented with symptoms such as right upper quadrant abdominal pain or headache with visual disturbances or PE-related findings (low platelets, elevated liver transaminases, Vascular Fetal Growth Restriction)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Biomarkers ratio | Every day from date of inclusion until date of delivery or up to 21 days whichever came first, in women with severe preeclampsia
  sFlt-1/PlGF ratio

SECONDARY OUTCOMES:
Biomarkers ratio | Every two day from date of inclusion until date of delivery or up to 21 days whichever came first, in women with moderate preeclampsia
  sFlt-1/PlGF ratio
Biomarkers ratio | Weekly from date of inclusion until date of delivery or up to 3 weeks whichever came first, in women with mild preeclampsia
  sFlt-1/PlGF ratio
Maternal outcome | From date of inclusion until the date of first documented event, assessed up to 24 weeks
  Incidence of retroplacental hematoma, or HELLP syndrome (Hemolysis, Elevated liver enzyme levels, and Low Platelet levels), or Renal failure.
Fetal outcome | From date of inclusion until the date of first documented event, assessed up to 24 weeks
  Incidence of a composite fetal outcome (in utero fetal death or, Intrauterine growth restriction, or APGAR < 7, or Prematurity)
Fetal outcome | Date of delivery
  Rate of in utero fetal death or, Intrauterine growth restriction, or APGAR < 7, or Prematurity

CONTACTS AND LOCATIONS:
Overall Officials: Dalenda Chelli, MD, Study Chair — Maternité de la Rabta - Tunis; Youcef Djedid, MD, Principal Investigator — Maternité de la Rabta - Tunis
Locations (1):
- Maternity Center of Tunis, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No